CLINICAL TRIAL: NCT02177877
Title: A Biosensor for Tracking Seizures: Linking a Wrist Accelerometer to an Online Epilepsy Diary
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: SmartMonitor (Unknown)
Responsible Party: Principal Investigator, Scheherazade Le, Principle Investigator, Stanford University
Other Study IDs: SM-29027
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizures; Wrist accelerometer; Epilepsy diary; Seizure detection; Biosensor
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will assess whether a movement detecting wristwatch can accurately detect seizures and seizure characteristics and record them into an online epilepsy diary. The patients may manually record a description into the online epilepsy diary of the symptoms they experienced before, during or after the seizure.

DETAILED DESCRIPTION:
Typically, health care providers receive inaccurate patient self- reports. This pilot trial will document the feasibility of accurately recording and logging seizures into a cloud-based diary, under circumstances of controlled video-EEG monitoring to serve as a comparison "gold standard." More explicitly, we are testing the efficacy of the wristwatch in capturing movement parameters correlated with seizure activity and whether these parameters can be accurately uploaded into an online epilepsy diary. In the future, biosensor data could be valuable to more precisely obtain seizure data for clinical decision making as well as use in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

-Adults over the age of 18 with known epileptic convulsive seizures already being admitted to the EMU for continuous video EEG.

Exclusion Criteria:

* Patients with only non-convulsive events or only psychogenic non-epileptic seizures.
* Patients who are unable to provide consent.
* Patients who have developmental delay.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with epilepsy over the age of 18 enrolled at the Stanford Epilepsy Monitoring Unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Capture rate of convulsive seizure events by the watch and watch-diary interface compared to video electroencephalography (vEEG) | up to 7 days

SECONDARY OUTCOMES:
Capture rate of non-seizure events by the watch and watch-diary interface compared to vEEG | up to 7 days
Frequency of movements of the watch diary interface vs vEEG | up to 7 days
Amplitude of movements of the watch diary interface vs vEEG | up to 7 days
Seizure semiology captured by the watch vs vEEG. | up to 7 days.
Specificity of audio recordings of the watch vs vEEG | up to 7 days
  Will record audio through the watch and vEEG to assess the specificity of this parameter for epileptic vs nonepileptic seizures

OTHER OUTCOMES:
Recording accuracy of convulsive seizure events by the watch and watch-diary interface compared to vEEG | up to 7 days
  Will measure the date and time, duration and shake intensity of convulsive seizure events by the watch and watch-diary interface compared to vEEG
Feasibility of use of device | up to 7 days
  Will survey whether the device was easy, neutral, difficult to use
Recording accuracy of partial seizures | up to 7 days
  Will compare partial seizure events detected by vEEG vs. watch-diary vs. patient log vs. caregiver log

CONTACTS AND LOCATIONS:
Overall Officials: Scheherazade Le, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

REFERENCES:
- [Result] Velez M, Fisher RS, Bartlett V, Le S. Tracking generalized tonic-clonic seizures with a wrist accelerometer linked to an online database. Seizure. 2016 Jul;39:13-18. doi: 10.1016/j.seizure.2016.04.009. Epub 2016 Apr 29. PMID 27205871